CLINICAL TRIAL: NCT03013387
Title: Phase II, Dosimetry-Guided, Peptide Receptor Radiotherapy (PRRT) With 90Y-DOTA- tyr3-Octreotide (90Y-DOTATOC) in Children and Adults With Neuroendocrine and Other Somatostatin Receptor Expressing Tumors
Brief Title: Dosimetry Guided PRRT With 90Y-DOTATOC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This project has undergone a significant amount of updates and has been resubmitted under IRB# 201708778
Sponsor: Sue O'Dorisio (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Sue O'Dorisio, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201611818; 1R01CA167632-01 (NIH)
Record Dates: First submitted 2016-12-14; First posted 2017-01-06 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Neuroendrocrine Tumors; Meningioma; Neuroblastoma; Medulloblastoma
MeSH Terms: conditions — Meningioma; Neuroblastoma; Medulloblastoma | interventions — 90Y-octreotide, DOTA-Tyr(3)-; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Whole Body Imaging; Amino Acids; arginyllysine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRRT with 90Y--DOTA-tyr3-Octreotide (Experimental): The 90Y--DOTA-tyr3-Octreotide initial, Cycle 1 dose will be 50 mCi/m2 in children; 120 mCi in adults. Treatment consists of 3 cycles, 6-8 weeks apart. Cycle 1 dose is fixed. Cycles 2 and 3 doses will be determined by dosimetry-based calculation of renal doses from previous cycles; total renal dose ≤ 23Gy. 90Y-DOTA-tyr3-Octreotide will be administered with an amino acid solution to prevent radiation damage to kidneys. Amino acid infusion will begin 30 min prior to infusion of 90Y-DOTATOC and continue 3.5 hrs after infusion of study drugs.
  68Ga-DOTATOC will be administered intravenously to perform the PET/CT scan. The dose will be 3-5 mCi (target 4mCi). The pediatric dose will be 0.043 mCi/kg with a minimum dose of 0.3 mCi and a maximum dose of 3 mCi in children <18 years old.
  Interventions: Radiation: 90Y-DOTA-3-tyr-Octreotide; Procedure: Positron Emission Tomography (PET) whole body scan; Drug: Amino Acids

INTERVENTIONS:
Radiation: 90Y-DOTA-3-tyr-Octreotide — 90Y-DOTATOC is a radiopharmaceutical that will be used l as a treatment for both children and adults with neuroendocrine and other somatostatin receptor positive tumors.
  Other Names: 90Y-DOTATOC
Procedure: Positron Emission Tomography (PET) whole body scan — 68Ga-DOTATOC is a radiopharmaceutical used in PET scans to identify tumors as it can adhere to Somatostatin Receptors.
  Other Names: 68Ga-DOTATOC PET
Drug: Amino Acids — This is a solution of amino acids that will decrease the amount of 90Y-DOTATOC that recirculates through the body after injection, therefore decreasing radiation dose to the kidneys.
  Other Names: Lysine and Arginine

SUMMARY:
This is a Phase 2 peptide receptor radionuclide therapy trial of 90Y-DOTATOC in patients with somatostatin receptor positive tumors.

DETAILED DESCRIPTION:
This is a Phase 2 peptide receptor radionuclide therapy trial of 90Y-DOTATOC in patients with somatostatin receptor positive tumors. The somatostatin receptor targeting of the therapeutic will be checked with 68Ga-DOTATOC PET-CT imaging prior to therapy. Treatment consists of 3 cycles, 6-8 weeks apart. Cycle 1 dose is fixed with Cycles 2 and 3 doses to be determined by dosimetry-based calculation of renal doses from previous cycles not to exceed 23 Gy for the total renal dose.

The goals of the project are to

1. Demonstrate safety and efficacy of renal uptake dosimetry-guided peptide receptor radiotherapy (PRRT) using 90Y-DOTA-tyr3-Octreotide (90Y-DOTATOC) in patients with neuroendocrine and other somatostatin receptor expressing tumors.
2. Monitor all adverse events associated with peptide receptor radiotherapy using 90Y-DOTATOC.
3. Establish 68Ga-DOTA-tyr3-Octreotide (68Ga-DOTATOC) PET/CT as an accurate technique for diagnosis, staging, treatment targeting, and monitoring response to 90Y-DOTATOC therapy.

ELIGIBILITY:
Inclusion Criteria

1. Disease not amenable to standard treatment (nonresectable or disease present after one or more surgeries and/or Sandostatin treatment) or subject has failed existing first line chemotherapy, biologic therapy, targeted agent therapy or radiation therapy.
2. Participation in Iowa Neuroendocrine Tumor Registry.
3. A pathologically confirmed (histology or cytology) malignant neoplasm with at least one target lesion that is confirmed by conventional imaging (CT or MRI) and is determined to express somatostatin receptors by 68Ga-DOTATOC (TATE) PET within 120 days prior to entry into the trial.
4. The target lesion is one that either has never received external beam radiation or has been previously irradiated and has since demonstrated progression. Any local irradiation of the target lesion or any non-target lesions via external beam, conformal or stereotactic radiation treatments must have occurred more than 4 weeks prior to study drug administration. Any full cranial-spinal radiation, whether or not a target lesion is included in the field, must have occurred more than 3 months prior to study drug administration.
5. Life expectancy > 2 months at the time of study drug administration.
6. Archival tissue from a previous biopsy will be required.
7. Age ≥ 6 months-90 years at the time of study drug administration.
8. Performance status as determined by Karnofsky ≥ 60 or Lansky Play Scale ≥ 60% at the time of study drug administration.
9. Completion of Norfolk Quality of Life Questionnaire.
10. Within 7-10 days of study drug administration, patients must have normal organ and marrow function as defined below:

    * absolute neutrophil count ≥1000/mm3
    * Platelets ≥90,000/mm3
    * total bilirubin <3X ULN for age
    * AST(SGOT) & ALT(SGPT) ≤10X institutional upper limit of normal for age
    * Urinalysis no greater than 1+ hematuria or proteinuria. Adults(age18 or >): Serum creatinine ≤ 1.2 mg/dl; if serum creatinine is >1.2 mg/dL,nuclear GFR will be measured. GFR will need to be ≥ 80 ml/min/1.73m2 for subjects ≤40 years old,
    * Renal function

      * 70 ml/min/1.73m2 for subjects between 41-50;
      * 60 ml/min/1.73m2 for subjects between 51-60;
      * 50 ml/min/1.73m2 for subjects > 60 years old. Children(age <18): nuclear GFR ≥ 80 mL/min/1.73 m2

        * Renal function criteria based on our previous experience with 90Y-DOTATOC therapy and known changes in GFR with age.
11. The effects of 90Y-DOTA-tyr3-Octreotide on the developing human fetus are unknown. For this reason and because Class C agents are known to be teratogenic, women and men of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
12. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

1. Pregnant women are excluded from this study because 90Y-DOTATOC is a Class C agent with potential teratogenic or abortifacient effects.
2. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 90Y-DOTATOC, breastfeeding should be discontinued until 6 weeks after the last administration of study drug.
3. Surgery within 4 weeks of study drug administration.
4. External beam radiation to both kidneys (scatter doses of <500 cGy to a single kidney or radiation to < 50% of a single kidney is acceptable).
5. Prior PRRT with 90Y-DOTATOC (TATE) or 177Lu-DOTATOC (TATE) or 131I-MIBG therapy for this malignancy.
6. Another investigational drug within 4 weeks of study drug administration.
7. Concurrent, malignant disease for which patient is on active therapy.
8. Another significant medical, psychiatric, or surgical condition which is currently uncontrolled by treatment and which would likely affect the subject's ability to complete this protocol.
9. Any subject for whom, in the opinion of their physician, a 12-hour discontinuation of somatostatin analogue therapy represents a health risk. Also subjects who have received long-acting somatostatin analogue in the past 28 days or long-acting lanreotide within the past 8 weeks are excluded. Subjects may be maintained on short acting octreotide during the time from last injection of long-acting somatostatin analogue until 12 hrs prior to injection of study drug. Known antibodies to Octreotide, Lanreotide, or DOTATOC or history of allergic reactions attributed to compounds of similar chemical or biologic composition to 90Y-DOTATOC.
10. Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) of study drug administration or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
11. Uncontrolled illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Subject weighs more than 450 pounds. (Subjects who weigh more than 450 pounds will not be able to fit inside the imaging machines.)
13. Inability to lie still for the entire imaging time (due to cough, severe arthritis, etc.)

Ages: 6 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy as assessed by change and defined as complete response, partial response or stable disease (CR+PR+SD) | Lesions will be quantified and compared between pre-therapy and through follow-up visits: 1) occurring 3-4 months after treatment 3 and 2) occurring 6-9 months after treatment 3
  Tumor response defined according to RECIST1.1 criteria applied on up to five target lesions (primary tumor, up to two: liver lesions, nodal metastases, and a metastatic lesion in other organs) that will be quantified and compared between pre-therapy and 3-9 months post-therapy high-resolution, contrast-enhanced CTs. 90Y-DOTATOC will be deemed worthy of further study if its associated response rate is ≥ 0.60, and clinically uninteresting if its rate is ≤ 0.40. Enrollment will proceed according to an optimal Simon two-stage study design. Sixteen (16) enrolled in the first stage; if 7 or fewer patients respond, the arm will be closed and the treatment ruled clinically uninteresting. Otherwise, an additional 30 will be enrolled. If 24 or more responses are observed in the total of 46 subjects, then the treatment will be ruled worthy. The study design has a probability of early termination equal to 0.72. Power to detect efficacy is 0.80 with a type 1 error rate of 0.05.
Renal, hematologic, and clinical toxicities | Lesions will be quantified and compared between pre-therapy and through follow-up visits: 1) occurring 3-4 months after treatment 3 and 2) occurring 6-9 months after treatment 3
  Adverse events will be recorded and reported in tabular form by type and grade. If four or more subjects experience renal toxicity ≥ Grade 4, the radiopharmaceutical will be declared too toxic and the trial will be stopped. If any other irreversible Grade 4 toxicity is observed in four or more subjects, the treatment will be declared too toxic and will be stopped. Adverse events will be graded according to the most recent CTE guidelines.

SECONDARY OUTCOMES:
Determine response to therapy of lesions identified by 68Ga-DOTATOC PET/CT but not identified on Octreoscan as a confirmatory measure of true positivity of the Ga-68 DOTATOC avid lesion | Lesions will be quantified and compared between pre-therapy and through follow-up visits: 1) occurring 3-4 months after treatment 3 and 2) occurring 6-9 months after treatment 3
  For subjects who participated in the 68Ga-DOTATOC Comparator trial (IRB # 201212736), the number, size, and location of discordant lesions between 68Ga-DOTATOC PET/CT and Octreoscan will have been tabulated. This analysis will be updated using the results of post- therapy 68Ga-DOTATOC PET/CT for those patients who participated in the comparator study, but only received the initial 68Ga-DOTATOC PET/CT due to progression on the Octreoscan + high-resolution, contrast-enhanced CT. Lesions that were positive on PET, but negative on Octreoscan will be considered true positive if a response to PRRT is documented after either Cycle 1 or at 6-9 month followup following last 90Y-DOTATOC infusion.
  For subjects who did not participate in the 68Ga-DOTATOC Comparator trial, all 68Ga-DOTATOC PET/CT scans will be acquired as part of this study; number, size, and location of lesions will be analyzed between first and subsequent 68Ga-DOTATOC PET/CTs.
Determine if Standard Uptake Value (SUV) on initial 68Ga-DOTATOC PET imaging correlates with SSTR2 expression as measured by quantitative messenger RNA (qPCR) or immunohistochemistry (IHC) on the diagnostic biopsy specimen | Lesions will be quantified and compared between pre-therapy and through follow-up visits: 1) occurring 3-4 months after treatment 3 and 2) occurring 6-9 months after treatment 3
  Compare maximum SUVs of primary tumor, liver lesions, and extra-hepatic lesions with expression level of sst2 RNA and IHC on fresh frozen tissue, or paraffin embedded samples (block(s) or 10 unstained slides) to determine whether or not any correlation exists between SUVmax, sst2 expression, or sst2 protein and response to PRRT. The study is expected to delineate whether measurement of sst2 expression by either qRT-PCT or immunohistochemistry at diagnosis can predict response to 90Y-DOTATOC. We will construct a table tabulating SUVmax, level of RNA expression, and IHC level for all lesions biopsied. With 64 subjects the correlation between SUV max, RNA expression and IHC will be determined. Analysis of SUVmax compared with sst2 RNA and receptor protein expression on primary tumor and metastatic lesions will be considered worthy of further study if > 50% of lesions demonstrate a positive correlation.

CONTACTS AND LOCATIONS:
Overall Officials: M S O'Dorisio, MD, PhD, Principal Investigator — University of Iowa

IPD SHARING:
Plan to Share IPD: No